CLINICAL TRIAL: NCT01456754
Title: Effect of Feeding Frequency on Glucose and Insulin Metabolism and Substrate Partitioning in Impaired Glucose Tolerant (IGT) Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Nederlandse Zuivel Organisatie (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: MEC 10-3-057
Record Dates: First submitted 2011-09-26; First posted 2011-10-21 (Estimated); Last update posted 2011-12-15 (Estimated); Status verified 2011-12

CONDITIONS: Glucose Intolerance
Keywords: Insulin Metabolism; Glucose Metabolism; Substrate Partitioning; Muscle Biopsies; Feeding Frequency; Insulin
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High feeding frequency (14x) (Experimental)
  Interventions: Dietary Supplement: High feeding frequency (14x)
- low feeding frequency (3x) (Experimental)
  Interventions: Dietary Supplement: low feeding frequency (3x)

INTERVENTIONS:
Dietary Supplement: low feeding frequency (3x) — 3 meals a day
  Arms: low feeding frequency (3x)
Dietary Supplement: High feeding frequency (14x) — 14 meals a day
  Arms: High feeding frequency (14x)

SUMMARY:
The purpose of this study is to determine the effect of feeding frequency on glucose and insulin metabolism and substrate partitioning in impaired glucose tolerant (IGT) men.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 20-35 kg/m2
* Gender: Male
* Age: subjects has to be older than 18 and younger than 70 years old
* Impaired Glucose Tolerant (IGT) = plasma glucose, two hours after consuming 75g glucose, appears to be superior to 7.8mmol/l (normal level) but remains inferior to 11.1mmol/l (diabetes level) and fasting plasma glucose is less than 7.0mmol/l.
* Caucasian

Exclusion Criteria:

1. Lactose intolerant
2. Diabetes Mellitus
3. Cardiovascular diseases
4. Stomach and intestinal diseases
5. Normal glucose levels after 2 hours
6. Anticoagulants
7. Medication that has a effect on energy and glucose homeostasis and absorption of foods
8. Conditions or situations when subjects can't lose 500 ml blood

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-12; Primary Completion 2011-09 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Glucose metabolism | 24 hour profile
Insulin metabolism | 24 hour profile

SECONDARY OUTCOMES:
Change in substrate partitioning (fat, carbohydrate and protein oxidation) between the two intervention diets | 24 hour profiles
Metabolic markers (FFA and TG metabolism) | 24 hour profile

CONTACTS AND LOCATIONS:
Overall Officials: Wim Saris, Prof. MD, Principal Investigator — Maastricht University
Locations (1):
- University of Maastricht, Maastricht, Netherlands